CLINICAL TRIAL: NCT00853086
Title: United Kingdom Haemophilia Centre Doctor's Organisation (UKHCDO) - Novo Nordisk Collaboration on NovoSeven® Post Marketing Follow-up Measures
Brief Title: Post-marketing Safety Surveillance of NovoSeven® in Patients With Haemophilia and Inhibitors by Means of the UK Haemophilia Database
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7HAEM-3537; U1111-1130-5940 (Other: WHO)
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — recombinant FVIIa

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: activated recombinant human factor VII

INTERVENTIONS:
Drug: activated recombinant human factor VII — Safety data collection in connection with the use of the drug NovoSeven® in daily clinical practice
  Other Names: NovoSeven®; rFVIIa; F7

SUMMARY:
This study is conducted in Europe. The purpose of this retrospective study is to collect additional safety information of patients with haemophilia and inhibitors who are treated with rFVIIa.

DETAILED DESCRIPTION:
Non-interventional, retrospective data collection on standard treatments of haemophilia A and B patients with inhibitors in the UK.

ELIGIBILITY:
Inclusion Criteria:

* All haemophilia A or B patients with inhibitors treated with NovoSeven are included

Exclusion Criteria:

* No exclusion criteria beyond the contraindications described in the approved product information text

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from speciality practice settings
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Quantify number of thrombotic events in patients treated with the currently recommended dose of 90 microgram/kg compared with higher rFVIIa dose levels up to 270 microgram/kg in relation to number of treatment episodes. | Assessments at 6 month intervals

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Crawley, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com